CLINICAL TRIAL: NCT02659137
Title: HV Electrophysiology Study In Transcatheter Aortic Valve Implantation Patients
Acronym: HESITATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: 152042
Record Dates: First submitted 2016-01-04; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Left Bundle Branch Block; Transcatheter Aortic Valve Replacement; Transcatheter Aortic Valve Implantation
Keywords: LBBB; TAVI
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: HV measurement — Electrophysiology (EP) study during the TAVI procedure
  Other Names: Electrophysiology study; His-catheter; His catheter; EP study

SUMMARY:
TAVI induced LBBB is a complication that occurs between 7 and 65 % of the cases, numbers that differ considerably between devices. There is an increased risk of progression to total AV-block at follow-up, with the risk of brady-arrhythmic death.

The aim of the study is to elucidate the anatomical location of the conduction pathology of a TAVI induced LBBB. This could impact valve design and placement and thereby reduce the number of new LBBB induced by TAVI in the future. Furthermore, finding predictors for progression to a high degree AV block in the follow-up (and thus an indication for permanent pacemaker) could improve management of post-operative conduction abnormalities and prevent the risk of brady-arrhythmic death.

DETAILED DESCRIPTION:
A prospective, single center, non-randomized pilot study in which patients will undergo an electrophysiology (EP) study during the TAVI procedure.

All patients eligible for inclusion will undergo an electrophysiology (EP) study during the TAVI procedure. For the purpose of EP measurements, a His-catheter will be placed at the beginning of the procedure and remain in the same location until the end of the procedure.

Continuous HV measurements will be collected, together with a continuous surface ECG, during the entire TAVI procedure. The different steps in TAVI procedure will be registered.

During the study, patients will undergo regular electrocardiographic examinations at the outpatient clinic (before implantation, after implantation, before discharge and after 6 weeks, 6 and 12 months post-implantation). These are part of the standard healthcare after the TAVI procedure.

The research protocol has been approved by the ethical committee (METC).

ELIGIBILITY:
Inclusion Criteria:

* All patients must provide written informed consent

Exclusion Criteria:

* Pre-existent LBBB
* Pre-existent sick sinus syndrome
* Pre-existent high-degree atrioventricular block
* Pre-existent permanent pacemaker
* Patients unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing implantation of a TAVI device in the Maastricht University Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Presence of a conduction disturbance in the His-bundle on occurence of a left bundle branch block on surface electrocardiogram by registering the HV-time in milli-seconds during the TAVI procedure. | 2 hours (from beginning to the end of TAVI procedure)
  Evaluate the location of a LBBB.

SECONDARY OUTCOMES:
Persistency and/or progression of a TAVI induced LBBB by registering the presence of a LBBB or a high degree AV block (second degree AV block or complete AV block) on surface electrocardiogram (ECG). | at 1 day before TAVI procure, at 1 hour after TAVI procedure, at discharge, at 6 weeks, at 6 months, at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands